CLINICAL TRIAL: NCT00320268
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled Phase III Study of the Efficacy and Safety of Quetiapine Fumarate Sustained-Release (SEROQUEL®) as Monotherapy in the Treatment of Patients With MDD
Brief Title: Safety & Efficacy Study of Quetiapine Fumarate (SEROQUEL®) vs. Placebo in Major Depressive Disorder
Acronym: MOONSTONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00001; Moonstone
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Quetiapine fumarate, sustained release; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate

SUMMARY:
This study is to evaluate that (SEROQUEL®) quetiapine sustained-release is efficacious and safe in the treatment of patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented clinical diagnosis of Major Depressive Disorder.
* Be able to understand and comply with the requirements of the study.
* Able to understand and provide written informed consent

Exclusion Criteria:

* Patients (female) must not be pregnant or lactating
* Current or past diagnosis of stroke or transient ischemic attack (TIA).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2006-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from randomization to Week 6 in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score

SECONDARY OUTCOMES:
Change from randomization to each assessment in the MADRS total score
MADRS response, defined as a ≥50% reduction from randomization in the MADRS total score at Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Art Lazarus, MD, Study Director — AstraZeneca
Locations (37):
- United States (37):
  - Research Site, Little Rock, Arkansas
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Oceanside, California
  - Research Site, Santa Ana, California
  - Research Site, Denver, Colorado
  - Research Site, Norwich, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Oak Brook, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Farmington Hills, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Clementon, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Norristown, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Bellevue, Washington
  - Research Site, Seattle, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Brown Deer, Wisconsin

REFERENCES:
- [Derived] McIntyre RS, Gorwood P, Thase ME, Liss C, Desai D, Chen J, Bauer M. Early Symptom Improvement as a Predictor of Response to Extended Release Quetiapine in Major Depressive Disorder. J Clin Psychopharmacol. 2015 Dec;35(6):706-10. doi: 10.1097/JCP.0000000000000416. PMID 26474010
- [Derived] Weisler R, Montgomery SA, Earley WR, Szamosi J, Eriksson H. Extended release quetiapine fumarate in patients with major depressive disorder: suicidality data from acute and maintenance studies. J Clin Psychiatry. 2014 May;75(5):520-7. doi: 10.4088/JCP.13m08624. PMID 24816198
- [Derived] Weisler R, McIntyre RS. The role of extended-release quetiapine fumarate monotherapy in the treatment of patients with major depressive disorder. Expert Rev Neurother. 2013 Nov;13(11):1161-82. doi: 10.1586/14737175.2013.846520. PMID 24175720
- [Derived] Clayton AH, Locklear JC, Svedsater H, McIntyre RS. Sexual functioning in patients with major depressive disorder in randomized placebo-controlled studies of extended release quetiapine fumarate. CNS Spectr. 2014 Apr;19(2):182-96. doi: 10.1017/S1092852913000631. Epub 2013 Sep 25. PMID 24067192
- [Derived] Trivedi MH, Bandelow B, Demyttenaere K, Papakostas GI, Szamosi J, Earley W, Eriksson H. Evaluation of the effects of extended release quetiapine fumarate monotherapy on sleep disturbance in patients with major depressive disorder: a pooled analysis of four randomized acute studies. Int J Neuropsychopharmacol. 2013 Sep;16(8):1733-44. doi: 10.1017/S146114571300028X. Epub 2013 May 14. PMID 23673347
- [Derived] Vieta E, Bauer M, Montgomery S, McIntyre RS, Szamosi J, Earley WR, Eriksson H. Pooled analysis of sustained response rates for extended release quetiapine fumarate as monotherapy or adjunct to antidepressant therapy in patients with major depressive disorder. J Affect Disord. 2013 Sep 5;150(2):639-43. doi: 10.1016/j.jad.2013.01.052. Epub 2013 Mar 14. PMID 23497790
- [Derived] Thase ME, Montgomery S, Papakostas GI, Bauer M, Trivedi MH, Svedsater H, Locklear JC, Gustafsson U, Datto C, Eriksson H. Quetiapine XR monotherapy in major depressive disorder: a pooled analysis to assess the influence of baseline severity on efficacy. Int Clin Psychopharmacol. 2013 May;28(3):113-20. doi: 10.1097/YIC.0b013e32835fb971. PMID 23485955
- [Derived] Weisler RH, Montgomery SA, Earley WR, Szamosi J, Lazarus A. Efficacy of extended release quetiapine fumarate monotherapy in patients with major depressive disorder: a pooled analysis of two 6-week, double-blind, placebo-controlled studies. Int Clin Psychopharmacol. 2012 Jan;27(1):27-39. doi: 10.1097/YIC.0b013e32834d6f91. PMID 22027845
- [Derived] Weisler R, Joyce M, McGill L, Lazarus A, Szamosi J, Eriksson H; Moonstone Study Group. Extended release quetiapine fumarate monotherapy for major depressive disorder: results of a double-blind, randomized, placebo-controlled study. CNS Spectr. 2009 Jun;14(6):299-313. doi: 10.1017/s1092852900020307. PMID 19668121